CLINICAL TRIAL: NCT06114381
Title: Impact of Home Based Physical Exercise and Diet Management on Functional Performance and Depression Among Vitamin D Deficient Females
Brief Title: Physical Exercise and Diet Management in Vitamin D Deficient Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Mina Atef Georgui Elias, Lecturer, Department of Physical Therapy for Internal Medicine and Geriatrics, Faculty of Physical Therapy, Badr University in Cairo, Egypt., Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUC-IACUC-231015-43
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Home Based Physical Exercise (Experimental): This group composed of 30 participants who will receive full body physical exercise 6 days per week in addition to sun exposure as well as their vitamin D supplement for 6 weeks.
  Interventions: Other: Home Based Physical Exercise; Dietary Supplement: Vitamin D3 Supplements; Behavioral: Sun Exposure
- Diet management group (Experimental): This group composed of 30 participants who will receive dietary management and sun exposure as well as their vitamin D supplement for 6 weeks.
  Interventions: Dietary Supplement: Vitamin D3 Supplements; Other: Diet Management; Behavioral: Sun Exposure
- Sun Exposure and supplements (Experimental): This group composed of 30 participants who will receive only sun exposure as well as their vitamin D supplement for 6 weeks.
  Interventions: Dietary Supplement: Vitamin D3 Supplements; Behavioral: Sun Exposure
- Control group (No Intervention): This group composed of 30 participants who didn't receive any intervention

INTERVENTIONS:
Other: Home Based Physical Exercise — Home Exercise protocol consists of one hour divided to 3 minutes warm up",9 minutes' full body (lower limbs, abdomen, back and upper limbs) exercise composed of (aerobic and strengthening) and 3 minutes cool down 4 times per day and 15 minutes for each session 6 days with one day recovery and, with every day follow up with each patient to ensure they did the whole sets and instructed them the ways to each exercise, The total duration was 36 sessions (6 weeks) for each patient. Daily communication with all subjects through sending mobile messages 3 times every day. The message was to remind the participants and confirmation of their response.
  Arms: Home Based Physical Exercise
Dietary Supplement: Vitamin D3 Supplements — Vitamin D3 supplement (400mg) once daily.
  Arms: Diet management group; Home Based Physical Exercise; Sun Exposure and supplements
Other: Diet Management — Patients receive weekly diet program contains dietary sources of Vitamin D such as yolk eggs, tuna and milk.
  Arms: Diet management group
Behavioral: Sun Exposure — Patients regular exposure to sun once a day 30 minutes of sun exposure, between 10 a.m. and 4 p.m. daily. Exposure to the face, arms, hands, and legs without sunscreen
  Arms: Diet management group; Home Based Physical Exercise; Sun Exposure and supplements

SUMMARY:
The purpose of this study was to determine if home based physical exercises protocol and Diet management has an effect on functional performance and depression level related to vitamin D deficiency in females.

DETAILED DESCRIPTION:
This is a randomized controlled trial to study the effect of home based physical exercises in comparison to Diet management, sun exposure and vitamin D supplements on functional performance and depression level in females with vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose age ranged from 19-25 years.
* All participants have pre laboratory results with vitamin D deficiency less than 25 nmol/L and have been lasted for 6 months
* All participated subjects were female studying at Al-Jouf university, Al- Qurrayyat-Female Branch.

Exclusion Criteria:

* Chronic illness, liver, renal endocrine or autoimmune diseases.
* Patients who suffered from any cardiopulmonary diseases.
* History of fractures or any neuro-musculoskeletal disorders.

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Vitamin D3 blood test | 6 weeks
  Measuring of Vitamin D3 in Blood through lab test

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) | 6 weeks
  Depression questionnaire The HDRS (also known as the Ham-D) is the most widely used clinician-administered depression assessment scale. The original version contains 17 items (HDRS 17) pertaining to symptoms of depression experienced.
  The patients were brought and explained to them the method of the questionnaire, and then they answered all 17 questions and the numbers for each patient were collected and written down.
6 Minutes Walk Test | 6 weeks
  Measuring the distance patient walked in 6 minutes (6 Minute walk distance)
Dyspnea Borg scale | 6 weeks
  t uses a scale from 0 to 10, where 0 represents no dyspnea and 10 represents maximal dyspnea. Scores are obtained at the end of the 6MWD test and reflect the maximum degree of dyspnea at any time during the walk.

CONTACTS AND LOCATIONS:
Overall Officials: Wael OA Abd El-Khalek, Dr., Study Chair — Dept of Basic Sciences, Faculty of PT, BUC, Cairo, Egypt.; Doaa Saeed, Dr., Study Chair — Dept of PT for women's health, Faculty of PT, BUC, Cairo, Egypt.; Mina AG Elias, Dr., Study Chair — Dept of PT for Internal Medicine & Geriatrics, Faculty of PT, BUC, Cairo, Egypt.; Heba A Bahey El-Deen, Prof. Dr., Principal Investigator — Dept of PT & Health Rehabilitation, College of Applied Medical Sciences, Jouf University, KSA.
Locations (1):
- College of Applied Medical Sciences, Jouf University, Kingdom of Saudi Arabia, Jazan, Al Jawf Region, Saudi Arabia